CLINICAL TRIAL: NCT07236476
Title: A Multicentre, Open-label, Dose-finding, Phase 2 Study to Investigate the Efficacy, and Safety of Different Doses of LY01021 in Controlled Ovarian Hyperstimulation(COH) for Female Subjects Undergoing Assisted Reproductive Technology (ART)
Brief Title: Identify Effective Doses of LY01021 in Controlled Ovarian Hyperstimulation (COH) for Female Subjects Undergoing Assisted Reproductive Technology (ART)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LY01021/CT-CHN-204
Record Dates: First submitted 2025-08-27; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Assisted Reproduction
Keywords: Controlled Ovarian Hyperstimulation (COH); Assisted Reproductive Technology (ART)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LY01021 (Experimental): Treatment group 40mg: oral LY01021; 40mg QD p.o.; Treatment group 30mg: oral LY01021; 30mg QD p.o.; Treatment group 20mg: oral LY01021; 20mg QD p.o.;
  Interventions: Drug: LY01021

INTERVENTIONS:
Drug: LY01021 — LY01021 should be taken orally once a day.

SUMMARY:
This is a multicentre, open-label, dose-finding, phase 2 study that will recruit approximately 90 female subjects undergoing COH for in vitro fertilization (IVF) or intracytoplasmic single sperm injection (ICSI). Three LY01021 dose groups of 40 mg QD, 30 mg QD, and 20 mg QD will be included, with not exceed 45 subjects in each group to investigate the efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent of subjects and their spouses;
* Married infertile female subjects aged 20 to 40 years (40 years exclusive) with indications for in vitro fertilization-embryo transfer (IVF-ET) or intracytoplasmic sperm injection (ICSI);
* Weight 45Kg ~ 80Kg (both inclusive), and body mass index (BMI) 19.0 ~ 28.0kg/m2;
* Regular menstrual cycle (24 ~ 35 days, both inclusive) for the last 3 months prior to screening;
* Anticipated normal ovarian response;
* Willingness of the subject to undergo fresh cycle transfer with one or two embryos at a time in the first IVF-ET cycle；
* Normal cervical cytology results (TCT) or with limited clinically significance within 6 months prior to screening; or subjects with atypical squamous cells of undetermined significance (ASC-US) of TCT tested negative for high-risk types of human papillomavirus (HPV).

Exclusion Criteria:

* Prior to screening, individuals underwent three or more IVF/ICSI-ET COH cycles without achieving clinical pregnancy；
* Previous IVF/ ICSI failure due to sperm/fertilization problems/low fertilization rate(<30%) and no improvement in related medical condition;
* Subjects with more than 2 times of spontaneous abortion;
* Subjects at high risk of OHSS, judged by the investigator according to the Golan classification (e.g., those with moderate to severe OHSS during previous COH cycles, polycystic ovary syndrome (PCOS), or with previous cancelled COH cycles due to OHSS);
* Subjects with low ovarian function;
* Any pregnancy that occurred within 3 months prior to screening;
* Unexplained abnormal vaginal bleeding within 6 months prior to screening;
* Subjects with serious infection, severe trauma or major surgical procedure within 6 months prior to screening.
* ALT and AST levels at the screening visit or the start of ovarian stimulation were more than twice the upper limit of normal;
* Positive serum β-hCG test at the screening visit or the start day of ovarian stimulation;
* Past medical history or gynecological ultrasound indicates clinically significant conditions;
* Any disease or symptom that can affect systemic function or may affect the absorption, accumulation, metabolism, or excretion of the test drug (e.g., chronic intestinal diseases, Crohn's disease, ulcerative colitis).
* Major systemic diseases, endocrine or metabolic abnormalities;
* Thromboembolic diseases or a history of thromboembolic diseases;
* The subject or her spouse or both of them carry a chromosomal abnormality, or suffer from a known monogenic hereditary disease or a severe disease with genetic susceptibility requiring pre-implantation genetic testing (excluding chromosomal polymorphisms);
* Malignant tumor or history of malignant tumor (except basal cell or squamous cell skin cancer, papillary thyroid carcinoma, in situ cancer );
* Use of fertility regulators within 1 month prior to ovarian stimulation, such as clomiphene citrate, letrozole, gonadotropins (Gn), hormonal drugs (including oral contraceptives, estrogens, progestogens, etc.) bromocriptine, etc..
* Subjects who have used strong inducers/inhibitors of cytochrome P450 3A4 (CYP3A4), strong inducers/inhibitors of P-glycoprotein (P-gp), or gastric acid secretion inhibitors within 2 weeks or 5 half-lives (whichever is longer) before the first administration of LY01021;
* Any other reasons deemed by the researcher as unsuitable for participation in this study.

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Inhibition rate of premature LH surge | From Day 5 to the hCG injection 1 day

SECONDARY OUTCOMES:
Number of oocyte retrieved per COH cycle | On oocyte retrieval 1 day
2PN rate. | 16-18 hours (h) after fertilization
High quality embryo rate. | 3 days after fertilization
Chemical pregnancy rate. | 13-15 days after transplantation
Clinical pregnancy rate. | 30-37 days after transplantation
Persistent pregnancy rate. | 70-84 days after transplantation
Adverse events. | Through study completion, an average of 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No